CLINICAL TRIAL: NCT00249574
Title: HCV Treatment of IDUs After Buprenorphine Stabilization
Brief Title: Bridging Active Heroin Users to Hepatitis C Treatment Using Buprenorphine - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Organization to Achieve Solutions in Substance Abuse (OASIS) (Other)
Responsible Party: Diana Sylvestre, O.A.S.I.S
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15629-1; R01-15629-1
Expanded Access: Available
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2008-12

CONDITIONS: Hepatitis C; Heroin Dependence
Keywords: heroin addiction
MeSH Terms: conditions — Hepatitis C; Heroin Dependence | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pegInterferon (Experimental): Open label, observational trial to determine the safety of HCV treatment in active IDUs stabilized on buprenorphine/naloxone
  Interventions: Drug: Buprenorphine/naloxone; Drug: pegInterferon

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Human subjects HIV, HCV
Drug: pegInterferon — intervention drug 1. buprenorphine/naloxone. street-recruited heroin users induced on bup/naloxone for period of 3-6 months, after which the second intervention is offered. intervention drug 2: pegInterferon/ribavirin. subjects interested in initiation treatment for HCV are offered pegInterferon, 180ug SQ/wk and ribavirin, 800-1200 mg daily for the standard duration of HCV treatment as dictated by genotype.

SUMMARY:
The purpose of this study is to see whether street-recruited heroin users can be successfully treated for hepatitis C after stabilizing them on buprenorphine.

DETAILED DESCRIPTION:
This is a prospective pilot safety study based on the hypothesis that active, street-recruited heroin users can be successfully treated for hepatitis C after stabilization on buprenorphine. Eligible subjects will be actively using heroin and have hepatitis C viremia; screening will occur at street-based sites like syringe exchange programs. Those who are eligible will sign informed consent, and then be asked to attend 3 weekly educational sessions about hepatitis C and addiction as well as undergo an intake interview. After this, subjects will be inducted onto buprenorphine/naloxone combination therapy (Suboxone) and receive this medication for 12-24 weeks. Once reaching the 12-24 week study time point, subjects will have the option of a 12-week Suboxone taper, or instead of undergoing 6-12 months of hepatitis C treatment with pegylated interferon and ribavirin while being maintained on Suboxone. Once completing hepatitis C treatment, subjects will undergo a 24-week Suboxone taper, or be transitioned to outpatient Suboxone therapy by a medical provider.

ELIGIBILITY:
Inclusion Criteria:

* Active heroin or other illicit opioid use
* Active hepatitis C
* No medical or psychiatric contraindications
* Able to sign informed consent

Exclusion Criteria:

* No opiate dependence
* Age <18
* Unable or uninterested in attending weekly group sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety assessments

SECONDARY OUTCOMES:
Effectiveness of medication
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Sylvestre, M.D., Principal Investigator — Organization to Achieve Solutions in Substance Abuse (OASIS)
Locations (1):
- O.A.S.I.S., Oakland, California, United States